CLINICAL TRIAL: NCT06031155
Title: Swedish Esophageal and Cardia Cancer Study
Acronym: SECC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jesper Lagergren, Professor of Surgery, Karolinska Institutet
Other Study IDs: SECC
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Oesophageal Cancer; Surgery; Survivorship; Quality of Life
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of this nationwide Swedish project is to identify strategies that can help reduce the suffering and improve the survivorship among patients surgically treated for oesophageal cancer. This objective can be accomplished by a broad research approach that aims to:

1. describe health-related quality of life (HRQL)
2. identify risk factors and preventive actions for poor HRQL

DETAILED DESCRIPTION:
This is a Swedish nationwide, prospective, and population-based cohort including 90% of all patients operated on for esophageal or gastroesophageal junctional cancer in Sweden between 1st April 2001 and 31st December 2005. Detailed clinical data were continuously collected from medical records based on a predefined study protocol to ensure uniformity. The clinical data collected included patient and tumor characteristics, treatment details, and follow-up on complications. Patients were followed up with health-related quality of life (HRQL) questionnaires. The core questionnaire (EORTC QLQ-C30) was used to measure aspects of HRQL and symptoms that are applicable for cancer patient in general, whereas the esophageal cancer-specific module (EORTC QLQ-OES18) measured symptoms common among esophageal cancer patients. HRQL was assessed 6 months, 3, 5, 10 and 15 years after surgery while the 20-year follow-up is ongoing. All questionnaires were self-administered, delivered by mail and up to three reminders were sent if required. Collection of HRQL data was obtained anonymously (patients sent their answers to a central administration and not to the treating department). The all-cause and disease-specific mortality was assessed by linkage to the Causes of Death Registry. Informed consent was obtained from each participant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are alive and able to participate in the project 6 months following surgery for oesophageal cancer are eligible to participate in the study.

Exclusion Criteria:

* Patients with cognitive impairment, who are unable to complete the measures in Swedish or are too unwell to complete the assessment, are excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included patients having been curatively treated, including surgical resection (esophagectomy), for esophageal or gastroesophageal junctional cancer (adenocarcinoma or squamous cell carcinoma) between April 2, 2001 and December 31, 2005.
Sampling Method: Non-Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2001-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
General health-related quality of life (HRQL) | 6 months, 3, 5, 10,15 and 20 years
  The questionnaire used to measure general HRQL was the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). This 30-item cancer-specific questionnaire includes one global quality of life scale, five functional scales (physical, role, emotional, cognitive, and social function), three symptom scales (fatigue, nausea, and pain), and six single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The questionnaire scores were transformed into 0-100 scales. Higher scores in the global quality of life scale, functional scales, and HRQL summary score represent better HRQL or function, while higher scores in the symptom scales or items correspond to more symptoms. Missing data were handled according to the EORTC scoring manual.
Disease specific health-related quality of life (HRQL) | 6 months, 3, 5, 10,15 and 20 years
  The questionnaire used to measure general HRQL was the European Organisation for Research and Treatment of Cancer Quality of Life Oesophageal Cancer Module 18 questionnaire (EORTC QLQ-OES18). This is an 18-item well-validated questionnaire measuring esophageal cancer-specific symptoms. It comprises four multi-item scales (dysphagia, eating difficulties, reflux, and pain) and six single items (trouble swallowing saliva, choking when swallowing, dry mouth, trouble with taste, trouble with coughing, and trouble talking). The response alternatives make up a four-point Likert scale: [1] 'Not at all', [2] 'A little', [3] 'Quite a bit' and [4] 'Very much'. The responses were transformed into a score within the range of 0-100. High scores in scales and single items represent high level of symptoms. Missing data were handled according to the EORTC scoring manual.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Lagergren, PhD, Principal Investigator — Karolinska Institutet